CLINICAL TRIAL: NCT03025308
Title: A Multicenter, Open-label, Long Term Extension Study to Assess the Safety and Efficacy of Filgotinib in Subjects With Rheumatoid Arthritis
Brief Title: Long Term Extension Study to Assess the Safety and Efficacy of Filgotinib in Adults With Rheumatoid Arthritis
Acronym: FINCH 4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alfasigma S.p.A. (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-417-0304; 2016-003630-25 (EudraCT Number)
Record Dates: First submitted 2017-01-17; First posted 2017-01-19 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — GLPG0634

STUDY DESIGN:
Masking Description: This study was originally designed and initiated as a double-blind study but the study design will change to open-label following implementation of the protocol amendment # 4.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Blinded Phase: Filgotinib 200 mg (Experimental): Filgotinib 200 mg plus placebo to match (PTM) filgotinib 100 mg for up to 6 years
  Interventions: Drug: Filgotinib; Drug: Placebo to match filgotinib
- Blinded Phase: Filgotinib 100 mg (Experimental): Filgotinib 100 mg plus PTM filgotinib 200 mg for up to 6 years
  Interventions: Drug: Filgotinib; Drug: Placebo to match filgotinib
- Open Label Phase: Filgotinib 200 mg (Experimental): Filgotinib 200 mg for up to 6 years
  Interventions: Drug: Filgotinib
- Open Label Phase: Filgotinib 100 mg (Experimental): Filgotinib 100 mg for up to 6 years
  Interventions: Drug: Filgotinib

INTERVENTIONS:
Drug: Filgotinib — Tablet(s) administered orally once daily
  Other Names: GS-6034; GLPG0634
Drug: Placebo to match filgotinib — Tablet(s) administered orally once daily
  Arms: Blinded Phase: Filgotinib 100 mg; Blinded Phase: Filgotinib 200 mg

SUMMARY:
The primary objective of this study is to evaluate the long-term safety and tolerability of filgotinib in participants who have completed one of the parent studies of filgotinib in rheumatoid arthritis (RA).

ELIGIBILITY:
Key Inclusion Criteria:

* Males or females who may benefit from filgotinib as judged by the investigator AND who completed a Gilead sponsored filgotinib parent study for RA as outlined below:

  * Have completed GS-US-417-0301, GS-US-417-0302 or GS-US-417-0303 on study drug

    * OR
  * Have completed GS-US-417-0302 on standard of care therapy due to RA non-responder status
* Females of childbearing potential must have a negative pregnancy test prior to first dose of study drug in the long term extension (LTE)
* Females of childbearing potential who engage in heterosexual intercourse must agree to protocol-approved methods of contraception

Key Exclusion Criteria:

* Diagnosis of an autoimmune or inflammatory joint disease other than RA, which would put the participant at risk by participating in the study or would interfere with study assessments/data interpretation, per judgment of the investigator
* Known hypersensitivity to the study drug or its excipients
* Any medical condition which would put the participant at risk by participating in the study or would interfere with study assessments/data interpretation, per judgment of the investigator

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2731 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants Experiencing Adverse Events (AEs) | Up to 6 years
Proportion of Participants Experiencing Clinically Significant Laboratory Abnormalities | Up to 6 years

SECONDARY OUTCOMES:
Proportion of Participants Achieving American College of Rheumatology- N (ACR-N) Response in Each Arm | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Alfasigma Study Director, Study Director — Alfasigma S.p.A.
Locations (345):
- United States (72):
  - Rheumatology Associates of North Alabama, PC, Huntsville, Alabama
  - Arthrocare, Arthritis Care & Research PC, Gilbert, Arizona
  - Arizona Arthritis & Rheumatology Associates, P.C., Phoenix, Arizona
  - Arizona Arthritis & Rheumatology Associates, P.C., Tucson, Arizona
  - Medvin Clinical Research, Covina, California
  - C.V. Mehta M.D. Medical Corporation, Hemet, California
  - University of California San Diego (UCSD) - Perlman Ambulatory Clinic, La Jolla, California
  - Keck Medicine of USC- Division of Rheumatology, Los Angeles, California
  - Desert Medical Advances, Palm Desert, California
  - Stanford University Hospitals and Clinics (Immunology & Rheumatology), Palo Alto, California
  - C.V. Mehta Medical Corporation, Riverside, California
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - Desert Valley Medical Group, Victorville, California
  - Medvin Clinical Research, Whittier, California
  - AARDS Research, Inc., Aventura, Florida
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Omega Research Consultants, LLC, DeBary, Florida
  - University of Florida College of Medicine, Jacksonville - Rheumatology Research, Jacksonville, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - San Marcus Research Clinic, Inc., Miami Lakes, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Omega Research Consultants LLC, Orlando, Florida
  - IRIS Research and Development, LLC, Plantation, Florida
  - Jefrey D. Lieberman, MD, P.C., Decatur, Georgia
  - Springfield Clinic, Springfield, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Center For Arthritis and Osteoporosis, Elizabethtown, Kentucky
  - Bluegrass Community Research, Inc., Lexington, Kentucky
  - Klein & Associates, M.D., P.A., Cumberland, Maryland
  - Arthritis Treatment Center, Frederick, Maryland
  - Klein & Associates, M.D., P.A., Hagerstown, Maryland
  - The Center For Rheumatology And Bone Research, Wheaton, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Umass Memorial Medical Center- Memorial Campus, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Shores Rheumatology, PC, Saint Clair Shores, Michigan
  - St. Paul Rheumatology, PA, Eagan, Minnesota
  - Arthritis Associates, PLLC, Hattiesburg, Mississippi
  - North Mississippi Medical Clinics, Inc., Tupelo, Mississippi
  - Clayton Medical Research, P.C., St Louis, Missouri
  - Arthritis Consultants, Inc., St Louis, Missouri
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Arthritis & Osteoporosis Associates, Freehold, New Jersey
  - Ocean Rheumatology, PA, Toms River, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - NYU Langone Ambulatory Care Brooklyn Heights, Brooklyn, New York
  - Weill Cornell Physicians At Brooklyn Heights, Brooklyn, New York
  - Joint And Muscle Research Institute, Charlotte, North Carolina
  - Physicians East, PA, Greenville, North Carolina
  - PMG Research of Salisbury, Salisbury, North Carolina
  - Paramount Medical Research & Consulting, LLC, Middleburg Heights, Ohio
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - The Oklahoma Center For Arthritis Therapy & Research, Inc., Tulsa, Oklahoma
  - East Penn Rheumatology Associates, Bethlehem, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Arthritis Group, PC, Philadelphia, Pennsylvania
  - Clinical Research Center of Reading LLC, Wyomissing, Pennsylvania
  - PA Regional Center For Arthritis And Osteoporosis Research, Wyomissing, Pennsylvania
  - Articularis Healthcare Inc., dba Columbia Arthritis Center, PA, Columbia, South Carolina
  - Carolina Rheumatology & Neurology Assoc., PC, Myrtle Beach, South Carolina
  - Articularis Healthcare Group d/b/a ACME Research, Orangeburg, South Carolina
  - Articularis Healthcare Group d/b/a Low Country Rheumatology, Summerville, South Carolina
  - Ramesh C. Gupta, M.D., Memphis, Tennessee
  - Diagnostic Group, Beaumont, Texas
  - Trinity Universal Research Associates, Inc, Carrollton, Texas
  - Adriana Pop-Moody MD Clinic PA, Corpus Christi, Texas
  - Arthritis Centers Of Texas, Dallas, Texas
  - Southwest Rheumatology Research, LLC, Mesquite, Texas
  - Trinity Universal Research Associates, Inc, Plano, Texas
  - Arthritis & Osteoporosis Center of South Texas, San Antonio, Texas
- Argentina (11):
  - Ceim Investigaciones Medicas Srl, Ciudad Autonoma, Buenos Aires
  - CIMEL, Buenos Aires
  - Onganizacion Medica de Investigacion S.A (OMI), Ciudad Autonoma Buenos Aires
  - Mautalen Salud e Investigación, Ciudad Autonoma Buenos Aires
  - Consultorios Reumatológicos Pampa, Ciudad Autonoma de Buenos Aire
  - Investigaciones Reumatologicas Y Osteologicas (IRO) SRL, Ciudad Autonoma
  - Instituto De Reumatologia, Mendoza
  - Instituto Médico Cer, Quilmes
  - Instituto Iari, San Isidro
  - Cer San Juan, Centro Polivalente de Asistencia e Investigacion Clinica, San Juan
  - Centro Medico Privado de Reumatología, San Miguel de Tucumán
- Australia (3):
  - Rheumatology Research Unit, Maroochydore, Queensland
  - RK Will Pty Ltd, Victoria Park, Western Australia
  - Southern Clinical Research Pty Ltd, Hobart
- Belgium (4):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Reumaclinic Genk, Genk
  - Universitaire Ziekenhuizen (UZ) Leuven - Gasthuisberg, Leuven
  - Zna Jan Palfijn, Merksem
- Bulgaria (7):
  - "Medical Center Help" EOOD, Dobrich
  - "Medical Center- Hipokrat 2000" OOD, Haskovo
  - "UMHAT - Kaspela" EOOD, Plovdiv
  - "MHAT Lyulin" EAD, Department of Rheumatology, Sofia
  - Medical Center "N. I. Pirogov" EOOD, Sofia
  - "DCC Equita" EOOD, Varna
  - MHAT "Sveta Petka" AD, Department of Internal Diseases, Vidin
- Canada (2):
  - The Waterside Clinic, Barrie
  - Centre De Recherche Musculo Squelettique, Trois-Rivières
- Chile (3):
  - Quantum Research Santiago, Santiago
  - Someal SA, Santiago
  - Centro Medico De Reumatologia, Temuco
- Czechia (8):
  - MUDr. Michaela Blahova, revmatologicka ambulance s.r.o., Brno
  - L.K.N. Arthrocentrum, s.r.o., Hlučín
  - MUDr. Rosypalová, S.R.O., Ostrava-Poruba
  - Revmatologicky ustav, Prague
  - Revmatologicka Ambulance, Prague
  - Revmatologicka ambulance, Nuselska Poliklinika, Prague
  - Arthrocentrum spol.s.r.o., Prague Praha 10
  - Medical Plus, S.R.O., Uherské Hradiště
- Hôpital Lapeyronie, Service d'Immuno-Rhumatologic, Montpellier, France
- Germany (5):
  - Rheumapraxis Dr. med. Reiner Kurthen, Aachen
  - Schlosspark-Klinik, Berlin
  - Centrum f. inn. Diagn. und Therap. Rheumatologie/Immunologie, Frankfurt am Main
  - HRF II, Hamburger Rheuma Forsch. Zentrum II, MVZ f. Rheumatologie und Autoimmuned. Hamb. GmbH/ Dr. A. Everding GbR, Hamburg
  - Rheumazentrum Ratungen-Studienambulanz GbR, Ratingen
- Hong Kong (3):
  - Department of Medicine & Theraputics, The Chinese University of Hong Kong, Hong Kong
  - Department of Medicine, Queen Mary Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
- Hungary (8):
  - Betegapolo-Irgalmasrend Budai Irgalmasrendi Korhaz, Budapest
  - Revita Reumatológiai Kft., Budapest
  - Markhot Ferenc Oktatokorhaz es Rendelointezet; Reumatologiai Osztaly, Eger
  - Bekes Megyei Kozponti Korhaz, Pandy Kalman Tagkorhaz, Reumatologiai Osztaly, Gyula
  - Bacs Kiskun Megyei Korhaz Szedgedi Tudomanyegyetem Altalanos Orvostudomanyi Kar Oktatokorhaz Kalocsai Szent Kereszt Korh, Kalocsa
  - Pest Megyei Flor Ferenc Korhaz, Reumatologiai-es Fizioterapias Osztaly, Kistarcsa
  - Csongrad Megyei Dr. Bugyi Istvan Korhaz; Mozgasszervi Rehabilitacios Osztaly, Szentes
  - C-Med Rehabilitacios es Diagnosztikai Kozpont. Reumatologia, Székesfehérvár
- India (27):
  - Panchshil Hospital, Dep, Ahmedabad
  - B.J. Medical College and Civil Hospital, Ahmedabad
  - Chanre Rheumatology and Immunology Centre and Research, Bangalore
  - Chennai Meenakshi Multispeciality Hospital Ltd, Chennai
  - All India Institute of Medical Sciences, Delhi
  - Medanta - The Medicity, Gūrgaon
  - Gleneagles Global Hospitals, Hyderabad
  - Nizams Institute of Medical Sciences, Hyderabad
  - Shri Nidaan Hospital and Hope Fertility Centre, Jaipur
  - SR Kalla Memorial Gastro and General Hospital, Jaipur
  - Santokba Durlabhji Memorial Hospital Cum Medical Research Institute, Jaipur
  - Apollo Gleneagles Hospitals, Kolkata, Kolkata
  - Medical College & Hospital, Kolkata, Kolkata
  - Department of Rheumatology, KG Medical University, Lucknow
  - Kasturba Medical College Hospital, Mangalore
  - Vinaya Hospital and Research Centre, Mangalore
  - JSS Medical College and Hospital, Mysuru
  - Suretech Hospital and Research Centre Pvt Ltd, Nagpur
  - Maharaja Agrasen Hospital, New Delhi
  - Sir Ganga Ram Hospital, New Delhi
  - Centre for Rheumatic Disease, Hermes Doctor House, Pune
  - Deenanath Mangeshkar Hospital and Research Centre, Pune
  - Krishna Institute of Medical Sciences, Secunderabad
  - Rajiv Gandhi Institute of Medical Sciences and Government General Hospital, Srikakulam
  - Nirmal Hospital Private Limited, Surat
  - Medical College Baroda and Sir Sayajirao General Hospital, Vadodara
  - King George Hospital, Visakhapatnam
- St Vincent's University Hospital, Dublin, Ireland
- Israel (5):
  - Bnai Zion Medical Center, Haifa
  - The Lady Davis Carmel Medical Center, Haifa
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Medical Center, Tel Aviv
- Italy (2):
  - Departimento Cardio-toraco-vascolare Gestione delle Malattie Reumatiche e del Connettivo e Malattie Metaboliche dell'osso, Bologna, Bologna
  - Reumatologia, Milan
- Japan (56):
  - Chibaken Saiseikai Narashino Hospital, Narashino, Chiba
  - Medical Corporation Kojyokai Hirose Clinic, Tokorozawa, Saitama
  - Honjo Rheumatism Clinic, Takaoka, Toyama
  - Chiba University Hospital, Chiba
  - Kyushu Medical Center, Fukuoka
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Seirei Hamamatsu General Hospital, Hamamatsu
  - Hiroshima Rheumatology Clinic, Hiroshima
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital, Hiroshima
  - Hiroshima University Hospital, Hiroshima
  - Iizuka Hospital, Iizuka-shi
  - Saitama Medical University Hospital, Iruma-gun
  - Shimane University Hospital, Izumo
  - Kagoshima red cross hospital, Kagoshima
  - Matsubara Mayflower Hospital, Katō
  - Saitama Medical Center, Kawagoe
  - Hospital of the University of Occupational and Environmental Health, Japan, Kitakyushu-shi
  - Kobe University Hospital, Kobe
  - Kumamoto Orthopaedic Hospital, Kumamoto
  - Kurume University Medical Center, Kurume-shi
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - Kyoto University Hospital, Kyoto
  - Yu Family Clinic, Miyagi-gun
  - Zenjinkai Shiminnnomori Hospital, Miyazaki
  - Yoshida orthopaedic and rheumatology Clinic, Morioka
  - Nagaoka Red Cross Hospital, Nagaoka
  - Nagasaki Medical Hospital of Rheumatology, Nagasaki
  - Nagoya University Hospital, Nagoya
  - The Hospital of Hyogo College of Medine, Nishinomiya
  - Okayama Saiseikai General Hospital Outpatient Center, Okayama
  - Okayama University Hospital, Okayama
  - Ome Municipal General Hospital, Ōme
  - National Hospital Organization Sagamihara National Hospital, Sagamihara
  - Sanuki Municipal Hospital, Sanuki-shi
  - Sagawa Akira Rheumatology Clinic, Sapporo
  - Sapporo City General Hospital, Sapporo
  - Hokkaido University Hospital, Sapporo
  - Hokkaido Medical Center for Rheumatic Diseases, Sapporo
  - Sasebo Chuo Hospital, Sasebo-shi
  - Azuma Rheumatology Clinic, Sayama-shi
  - Niigata Rheumatic Center, Shibata
  - Shizuoka Welfare Hospital, Shizuoka
  - Osaka University Hospital, Suita-shi
  - Inoue Hospital, Takasaki-shi
  - St. Luke's International Hospital, Tokyo
  - Medical Corporation Uchida Clinic, Tokyo
  - Showa University East Hospital, Tokyo
  - Toho University Omori Medical Center, Tokyo
  - Toho University Ohashi Medical Center, Tokyo
  - Setagaya Rheumatic Clinic, Tokyo
  - Keio University Hospital, Tokyo
  - Teikyo University Hospital, Tokyo
  - Yuuai Medical Center, Tomigusuku-shi
  - University of Tsukuba Hospital, Tsukuba
  - Wakayama Medical University Hospital, Wakayama
  - Yokohama Minami Kyousai Hospital, Yokohama
- Malaysia (2):
  - Hospital Selayang, Batu Caves, Selangor
  - University Malaya Medical Centre, Kuala Lumpur
- Mexico (8):
  - Centro De Investigación Clínica De Morelia, Sc, Morelia, Michoacán
  - Kohler & Milstein Research S.A. de C.V., Mérida, Yucatán
  - Investigacion y Biomedicina de Chihuahua, S.C., Chihuahua City
  - Clinstile, S.A. De C.V., Mexico City
  - Clinosar Mexico. S.A. de C. V., Mexico City
  - Centro Peninsular De Investigacion Clinica S.C.P., Mérida
  - Biologicos Especializados, México
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey
- New Zealand (5):
  - Middlemore Clinical Trial, Papatoetoe, Auckland
  - Optimal Clinical Trials, Level 2, Auckland
  - Waikato Hospital, Hamilton
  - Clinical Trial Unit, CCHDB, Wellington Hospital, Newtown
  - Clinical Trials Unit, Timaru Hospital, Timaru
- Poland (19):
  - Gabinet Internistyczno-Reumatologiczny Piotr Adrian Klimiuk, Bialystok
  - Clinicmed, Bialystok
  - Szpital Uniwersytecki Nr 2, Klinka Reumatologii I Ukladowych Chorob Tkanki Lacznej, Bydgoszcz
  - Niepubliczny Zaklad Opieki Zdrowotnej BIF-MED S.C., Bytom
  - Nszoz Unica Cr, Dabrówka
  - Centrum Kliniczno-Badawcze J. Brzezicki, Elblag
  - Centrum Medyczne Pratia Gdynia, Gdynia
  - NZOZ Centrum Medyczna Sw. Lukasza w Kartuzach, Kartuzy
  - SILMEDIC Spolka z ograniczona odpowiedzialnoscia w Swindniku, Oddzial w Katowicach, Katowice
  - Nzoz Centrum Medyczne Promimed, Krakow
  - Twoja Przychodnia -Centrum Medyzcne Nowa Sol, Nowa Sól
  - Synexus Polska Sp. z.o.o. Oddzial w Porznaniu, Poznan
  - Centrum Badan Klinicznych S.C. Wieslawa Porawska, Lukasz Porawski, Poznan
  - Ai Centrum Medyczne, Poznan
  - Samodzielny Publiczny Zespol Opieki Zdrowotnej w Tomaszowie Lubelskim Lubelskim; Oddzial Reumatologiczy, Tomaszów Lubelski
  - Nasz Lekarz Przychodnie Medyczne, Torun
  - Reumatika -Centrum Reumatologii NZOZ, Warsaw
  - Centrum Medyczne AMED Warszawa Targówek, Warsaw
  - Centrum Medyczne Oporow, Wroclaw
- Romania (5):
  - Spitalul Judetean de Urgenta Bacau, Sectia Reumatologie, Bacau
  - S.C. Ianuli Med Consult S.R.L., Bucharest
  - Spitalul Clinic ,, Sf. Maria", Sectia Reumatologie, Bucharest
  - Spitalul Clinic,, Sf. Maria"", Departamentul de Medicina Interna si Reumatologie, Bucharest
  - Spitalul Clinic Judetean de Urgenta Tirgu Mures, Târgu Mureş
- Russia (15):
  - Territorial State Budgetary Healthcare Institution "Territorial Clinical Hospital", Barnaul
  - State Budgetary Healthcare Institution, Chelyabinsk Regional Clinical Hospital, Chelyabinsk
  - FSBEI of HE "Kazan State Medical University" of Ministry of Healthcare of the Russia Federation, Department of hospital therapy, Kazan'
  - Medical Center Maximum Zdorovia LLC, Kemerovo
  - Kemerovo State Medical University on the base of Regional Clinical Hospital for War Veterans, Kemerovo
  - Municipal Clinical Hospital No. 15 named after O.M. Filatov, Moscow
  - City Clinical Hospital #4 of Department of Healthcare of Moscow City, Moscow
  - M. Vladimirsky Moscow Regional Research Clinical Institute, Moscow
  - Municipal Clinical Hospital No. 40 Department of healthcare of Moscow City, Moscow
  - Nizhny Novgorod City Clinical Hospital #5, Nizhny Novgorod
  - Saint-Petersburg State Budgetary Healthcare Institution "Clinical rheumatology hospital # 25", Saint Petersburg
  - LLC Polyclinic of Private Security Personnel, Saint Petersburg
  - State Healthcare Institution, Regional Clinical Hospital, Saratov
  - LLC BioMed, Vladimir
  - State Autonomous Healthcare Institution of Yaroslavl region "Clinical Hospital for Emergency Medical Care n. a. N. V. Solovyev", Yaroslavl
- Serbia (4):
  - Institute Of Rheumatology, Belgrade
  - Military Medical Academy, Clinic of Rheumatology, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Institute For Treatment And Rehabilitation Niska Banja, Niška Banja
- Slovakia (3):
  - Neštátna Reumatologická Ambulancia, Bratislava
  - Reumex S.R.O., Rimavská Sobota
  - LERAM s.r.o., Topoľčany
- South Africa (5):
  - Arthritis Clinical Trial Centre, Cape Town
  - Netcare St. Augustine's Hospital, Durban
  - Umhlanga Netcare Medical Centre, Durban
  - Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg
  - Winelands Medical Research Centre, Stellenbosch
- South Korea (14):
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Daegu Catholic University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Eulji University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Inha University Hospital, Incheon
  - Chonbuk National University Medical School, Jeonju
  - Seoul National University Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Chung-Ang University Hospital Institutional Review Board, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
- Spain (9):
  - Complejo Hospitalario Universitario de Santiago, A Coruña
  - Hospital Universitario Cruces, Barakaldo
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Corporacio Santiaria Parc Tauli, Sabadell
  - Clínica Gaias, Santiago de Compostela
  - Hospital HM Nuestra Senora de la Esperanza, Santiago de Compostela
  - Hospital Clinico Universitario de Valencia, Valencia
- Taiwan (10):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital, Keelung, Keelung
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - Chi Mei Hospital, Chi Mei Medical Center, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Medical Foundation, Chang Gung Memorial Hospital, Linkou Branch, Taoyuan District
- Thailand (5):
  - Phramongkutklao Hospital, Division of Rheumatology, Department of Medicine, Bangkok
  - Rajavithi Hospital, Rheumatology and Allergy Unit, Bangkok
  - Faculty of Medicine Siriraj Hospital, Mahidol University, Division of Rheumatology, Department of Medicine, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Faculty of Medicine, Chiang Mai University, Chiang Mai
  - Faculty of Medicine, Prince of Songkla University, Songklanagarind Hospital, Songkhla
- Ukraine (19):
  - Municipal Institution Dnipropetrovsk 6th City Clinical Hospital of Dnipropetrovsk Regional Council, Dnipro
  - Municipal Nonprofit Enterprise of the Kharkiv Regional Council, Regional Hospital for War Veterans, Department of Therapy #1, Kharkiv
  - State Institution "National Institute of Therapy named after L.T. Maloyi" of National Academy of Medical Sciences of Ukraine", Kharkiv
  - Municipal Institution of Heath Care "Regional Clinical Hospital-Center Of Emergency Medicine & Disaster Medicine", Kharkiv
  - Municipal Nonprofit Enterprise "City Clinical Hospital #13" of the Kharkiv City Council, Department of Therapy, Kharkiv
  - Minicipal Institution "Kherson City Clinical Hospital n. a. Afanasiy and Olga Tropinykh", Department of Therapy #1, Kherson
  - Kyiv Oleksandrivska City Clinical Hospital, Department of Rheumatology # 2, Kyiv
  - Kyiv City Clinical Hospital #6, Department of Therapy, Kyiv
  - State Institution National Scientific Center M.D. Strazhesko Institute of Cardiology of NAMS of Ukraine, Kyiv
  - Municipal Institution of Kyiv Regional Council "Kyiv Regional Clinical Hospital", Highly Specialized Therapeutic Department, Kyiv
  - Lutsk City Clinical Hospital, Lutsk
  - Municipal Institution of Lviv Regional Council "Lviv Regional Clinical Hospital" Department of Rheumatology, Lviv
  - Municipal Nonprofit Enterprise "4-th City Clinical Hospital in Lviv", Department of Rheumatology, Lviv
  - Municipal Institution Odesa Regional Clinical Hospital, Polyclinic Department, Odesa
  - Vinnytsya Regional Clinical Hospital named after M. I. Pyrogova, Department of Rheumatology, Vinnytsia
  - City Clinical Hospital #1, Department of Rheumatology, Vinnytsia
  - Medical Centre Modern Clinic, LLC, Zaporizhzhya
  - Municipal Institution "City Hospital #1", Department of Therapy, Zaporizhzhya
  - Municipal Institution City Hospital #7, Department of Therapy, Zaporizhzhya
- United Kingdom (4):
  - NHS Lothian, Western General Hospital, Edinburgh
  - Princess Alexandra Hospital, Harlow
  - Northumbria Healthcare NHS Foundation Trust, North Shields
  - Warrington and Halton Hospitals Nhs Foundation Trust, Warrington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tanaka Y, Matsubara T, Atsumi T, Amano K, Ishiguro N, Hirata S, Yamaoka K, Combe BG, Nash P, Genovese M, Pechonkina A, Liu J, Kondo A, Fukada H, De Leonardis F, Takeuchi T. Safety and efficacy of filgotinib in Japanese patients with rheumatoid arthritis: Week 156 interim results in FINCH 4. Mod Rheumatol. 2025 Apr 8;35(3):425-433. doi: 10.1093/mr/roae099. PMID 39506562
- [Derived] Balsa A, Wassenberg S, Tanaka Y, Tournadre A, Orzechowski HD, Rajendran V, Lendl U, Stiers PJ, Watson C, Caporali R, Galloway J, Verschueren P. Effect of Filgotinib on Body Mass Index (BMI) and Effect of Baseline BMI on the Efficacy and Safety of Filgotinib in Rheumatoid Arthritis. Rheumatol Ther. 2023 Dec;10(6):1555-1574. doi: 10.1007/s40744-023-00599-1. Epub 2023 Sep 25. PMID 37747626
- [Derived] Combe B, Besuyen R, Gomez-Centeno A, Matsubara T, Sancho Jimenez JJ, Yin Z, Buch MH. Geographic Analysis of the Safety and Efficacy of Filgotinib in Rheumatoid Arthritis. Rheumatol Ther. 2023 Feb;10(1):35-51. doi: 10.1007/s40744-022-00494-1. Epub 2022 Oct 7. PMID 36205910